CLINICAL TRIAL: NCT05399979
Title: Fetal Heart Rate Changes and Labor Neuraxial Analgesia: a Machine Learning Approach
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Principal Investigator, Augusta University
Other Study IDs: 1567908
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Fetal Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Labor Neuraxial Analgesia — Labor Neuraxial Analgesia

SUMMARY:
This study aims to perform statistical inference and prediction of changes in fetal heart rate during active labor in healthy pregnant women by comparing three different machine learning methods

DETAILED DESCRIPTION:
Purpose: This study aims to perform statistical inference and prediction of changes in fetal heart rate during active labor in healthy pregnant women by comparing three different machine learning methods. Methods: A retrospective analysis of 1077 healthy laboring parturients receiving neuraxial analgesia was conducted. We compared a principal components regression model with treebased random forest, ridge regression, multiple regression, a general additive model, and elastic net in terms of prediction accuracy and interpretability for inference purposes.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Pregnancy requiring labor analgesia
* Active labor
* Request of neuraxial analgesia per patient and/or obstetrician
* Received combined spinal-epidural technique

Exclusion Criteria:

* Uterine tachysystole before neuraxial analgesia.
* Baseline blood pressure <90/60 mmHg.
* Third trimester hemorrhage
* Eclampsia
* Allergies to local anesthetics or fentanyl.
* Maternal fever.
* Pruritus before performance of neuraxial analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: -Pregnant patients admitted to the labor and delivery unit of an academic center
Sampling Method: Non-Probability Sample
Enrollment: 1077 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
fetal bradycardia | 15 minutes
  fetal heart rate under 120 lpm for more than 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University Medical Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No